CLINICAL TRIAL: NCT03182049
Title: Natural History of Granulomatosis With Polyangiitis: Clinical and Genetic Biomarkers of Airway Disease: North American Airway Collaborative (NoAAC) PR-03 Study
Brief Title: Natural History of Granulomatosis With Polyangiitis: Clinical and Genetic Biomarkers of Airway Disease NoAAC PR-03 Study
Acronym: NoAAC PR-03
Status: Withdrawn | Type: Observational
Why Stopped: Funding was not able to be secured for the study and no participants enrolled.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: North American Airway Collaborative (NoAAC) (Unknown); Vasculitis Patient Powered Research Network (VPPRN) (Unknown); Vasculitis Clinical Research Consortium (VCRC) (Network)
Responsible Party: Principal Investigator, Alexander Gelbard, MD, Assistant Professor, Department of Otolaryngology, Vanderbilt University Medical Center
Other Study IDs: 161780
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Granulomatosis With Polyangiitis
Keywords: GPA; Granulomatosis with polyangiitis; Wegener's granulomatosis; Subglottic Stenosis; Bronchial Stenosis
MeSH Terms: conditions — Granulomatosis with Polyangiitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We plan to obtain a small amount of blood at a time when other medically indicated labs, operative or office-based procedures occur.
  Excess tissue obtained at standard of care surgical biopsy will be preserved for molecular study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GPA (Wegener's granulomatosis) patients
  Interventions: Procedure: Airway assessment; Procedure: Rheumatology assessment

INTERVENTIONS:
Procedure: Airway assessment — Airway Specialist (Otolaryngology, Pulmonology, Thoracic Surgery), assess clinical location and degree of airway compromise, glottic mobility, and sinonasal disease.
Procedure: Rheumatology assessment — Clinically assess systemic function (renal/pulmonary ect), biochemical profile (routine labs), neurocognitive function, and completing entry BVAS tool.

SUMMARY:
The ultimate goal of this prospective natural history study is to define the natural history of the obstructive airway manifestations of Granulomatosis with polyangiitis (GPA).

Additionally this proposal seeks to develop biomarkers of disease activity and define their correlation with clinical outcomes in an effort to transform clinical care and shape future drug development for this devastating rare disease.

DETAILED DESCRIPTION:
Granulomatosis with polyangiitis (GPA, formerly known as Wegener's granulomatosis) is a rare multisystem necrotizing granulomatous vasculitis of small and medium vessels. Nearly 20% of GPA patients suffer life-threatening obstruction of their airways. Even when survived, airway involvement can render patients in this disease subset unable to communicate, struggling to breath, and dependent on a tracheostomy for survival. Airway disease frequently leads to irreversible physiologic impairment and is highly correlated with reduced quality of life in GPA.

Prior to the 1970s, patients with GPA had a 1-year mortality rate of >80%, primarily due to renal or lung failure. The introduction of combination cyclophosphamide and glucocorticoid treatment 4 decades ago greatly improved patient outcomes, turning this into a more chronic long-term disease. However, while progress has been made in the development of successful treatment regimes for systemic disease, the role of current therapies in ameliorating the airway complications of GPA is unknown. The evolution of GPA into a chronic disease has brought the management of the airway manifestations of GPA to the forefront. The natural history of the airway disease in GPA has never been longitudinally characterized, and there are no reliable biomarkers of clinical outcome.

In GPA the incidence of airway stenosis localized to the anatomic region below the vocal cord (subglottic stenosis) has been estimated to be 16%-50%. It may occur in isolation as the presenting symptom of GPA, or as a late-stage manifestation of disease. Although stenosis is frequently limited to the subglottis, it may extend up to involve to vocal cords, or down to involve the distal trachea and bronchi. Unfortunately, studies have documented a relatively high incidence of multilevel airway involvement (34%) in GPA. In one series of 44 patients, one in five had evidence of laryngeal stenosis. Studies have also found a high incidence of metachronous bronchial disease.

Laryngeal and Bronchial stenosis appear to be progressive and occur after the onset of subglottic stenosis, but the true natural history of airway involvement in GPA is unknown.

GPA is a member of the anti-neutrophil cytoplasmic antibody (ANCA) vasculitides. Given the strong association of GPA with ANCA production, much focus has been placed on understanding the mechanisms of ANCA production and pathogenesis. The factors by which ANCAs are initially generated are poorly understood. The majority of in vitro and animal model research implicating neutrophils and T cells as the principal inflammatory cells in GPA is surprising given the known impressive clinical treatment response to B cell depletion with rituximab. This discordance reinforces that the knowledge gap between pathogenesis and therapy is GPA is wide.

The distinction between focused airway disease and severe systemic disease has important therapeutic implications. The course of airway stenosis in GPA has been found to run independently of the systemic disease course and is often refractory to standard systemic therapy. In one representative case series, subglottic stenosis (SGS) was diagnosed in 49% of patients while they were receiving systemic treatment, and 56% of the patients who required tracheostomies did so despite having been treated for at least 2 months with systemic immunosuppressive agents. Developing novel therapeutics to control airway-focused GPA and prevent the development and/or progression of destructive airway damage is desperately needed.

Because of the small numbers of patients affected, and with clinical experience dispersed among a small number of clinical referral centers, the natural history of rare diseases is often poorly described. When knowledge about disease is insufficient to guide clinical development, well-designed natural history studies are critical to developing and proving the efficacy of novel therapeutics.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age.
* Stenotic Airway Disease (laryngeal, subglottic, distal tracheal or bronchial)

Exclusion Criteria:

* <18years of age
* Patients without capacity to consent for themselves
* History of significant laryngotracheal traumatic injury.
* Endotracheal intubation 2 years prior to presentation.
* Major anterior neck surgery.
* History of neck irradiation.
* History of caustic or thermal injury to the laryngotracheal complex.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Granulomtosis with Polyangiitis Population Affected by Obstructive Airway Disease patients are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Time to recurrent intervention (TTR) | 5 years
  The time between interventions aimed at preserving an open airway.

SECONDARY OUTCOMES:
Patient Reported Outcome Measures | 5 years
  Patient Quality of Life assessment: Voice (VHI10)
Patient Reported Outcome Measures | 5 years
  Patient Quality of Life assessment: Breathing (Clinical Dyspnea questionnaire or CDQ)
Patient Reported Outcome Measures | 5 years
  Patient Quality of Life assessment: Eating (EAT10)
Patient Reported Outcome Measures | 5 years
  Patient Quality of Life assessment: general quality of life (SF12)
Disease Assessment clinical tool | 5 years
  Birmingham Vasculitis Activity Score (BVAS)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Gelbard, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided